CLINICAL TRIAL: NCT06544603
Title: Effect of Laser Acupuncture for Traumatic Facial Paralysis: A Retrospective Study
Brief Title: Laser Acupuncture for Traumatic Facial Paralysis
Status: Completed | Type: Observational
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Laser-RS-2024
Record Dates: First submitted 2024-08-06; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-07

CONDITIONS: Traumatic Facial Paralysis
Keywords: traumatic facial paralysis; laser acupuncture; photobiomodulation; retrospective study
MeSH Terms: interventions — Lasers

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control group
- LA 3 month group: Laser acupuncture used a class IV Multiwave Locked System (MLS) laser (Mphi laser, ASA Srl, Vicenza, Italy). In LA group, we choose 5 acupoints on the affected side. It includes ST2(Si Bai), ST4(Di Cang), ST6(Jia Che), GB14(Yang Bai), GB20(Feng chi). We choose 6 acupoints, including LI4 (He Gu), LI11(Qu Chi), ST25 (Tian Shu), ST36 (Zu San Li), SP6 (San Yin Jiao), KI3 (Tai Xi), LR3 (Tai Chong).
  Laser acupuncture used have wavelength of 808 nm and 905nm, 1.2 W power (808nm is 1 W, 905 nm is 200 mW), continuous mode emission (808 nm) and pulsed mode emission (905 nm), 1500 Hz, 50% power level, 50% duty cycle, 8.35 J/cm2 dosimetry, 26.22 J for each point, 36 times total treatment.
  Interventions: Device: Multiwave Locked System (MLS) laser
- LA 6 month group: Laser acupuncture used a class IV Multiwave Locked System (MLS) laser (Mphi laser, ASA Srl, Vicenza, Italy). In LA group, we choose 5 acupoints on the affected side. It includes ST2(Si Bai), ST4(Di Cang), ST6(Jia Che), GB14(Yang Bai), GB20(Feng chi). We choose 6 acupoints, including LI4 (He Gu), LI11(Qu Chi), ST25 (Tian Shu), ST36 (Zu San Li), SP6 (San Yin Jiao), KI3 (Tai Xi), LR3 (Tai Chong).
  Laser acupuncture used have wavelength of 808 nm and 905nm, 1.2 W power (808nm is 1 W, 905 nm is 200 mW), continuous mode emission (808 nm) and pulsed mode emission (905 nm), 1500 Hz, 50% power level, 50% duty cycle, 8.35 J/cm2 dosimetry, 26.22 J for each point, 72 times total treatment.
  Interventions: Device: Multiwave Locked System (MLS) laser

INTERVENTIONS:
Device: Multiwave Locked System (MLS) laser — Laser probe directly contacts with skin of the all the acupoints. The probe was fixed on each point for 1 min. In this study, the laser acupuncture used have wavelength of 808 nm and 905nm, 1.2 W power (808nm is 1 W, 905 nm is 200 mW), continuous mode emission (808 nm) and pulsed mode emission (905 nm)
  Groups: LA 3 month group; LA 6 month group

SUMMARY:
Objective:

The objective of this study was to determine whether laser acupuncture therapy could relieve symptoms in patients with traumatic facial paralysis.

Methods:

This study was retrospective study including 174 patients that undergoing traumatic facial paralysis. All the patients received laser acupuncture (LA).

Patients were assigned to the LA 1 month group, LA 3 month group and LA 6 month group, with 58 patients in each group.

Clinical outcome measure comprised the House-Brackmann grading system, Facial Clinimetric Evaluation Scale (FaCE), Sunnybrook facial grading scale (SBFG), Facial Disability Index (FDI), electroneuronography (ENoG), electromyography (EMG) and Blink reflex

ELIGIBILITY:
Inclusion Criteria:

* 1, Patients diagnosed with traumatic facial paralysis 2, Patients were eligible if they were graded at House-Brackmann grade (HB) 3 or higher.

Exclusion Criteria:

- 1.Serious mental illness or social problems, and neurological disorders, and systemic diseases, such as malignant tumors, and other serious consumptive diseases.

2. Planning for pregnancy, those in pregnancy, or those who were lactating. 3. Neurotmesis by trauma.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enroll male and female participants aged 18-65 years, diagnosed with traumatic facial paralysis, with House-Brackmann grade (HB) 3 or higher.
  Exclusion criteria include serious mental illness or social problems, and neurological disorders, and systemic diseases, such as malignant tumors, and other serious consumptive diseases, planning for pregnancy, those in pregnancy, or those who were lactating, and neurotmesis by trauma.
  Participants will be recruited from outpatient clinics at Beijing Tongren Hospital through advertisements in the hospital and local community centers. All potential participants will undergo a thorough screening process, including a review of medical history and baseline tests, before providing written informed consent. Baseline characteristics will include age, gender, baseline HB, SB Grading, FaCE, ENoG, EMG and BR.
Sampling Method: Non-Probability Sample
Enrollment: 174 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-07-10 (Actual); Study Completion 2024-07-10 (Actual)

PRIMARY OUTCOMES:
House Brackmann Grading System (HB) | Baseline, month 3, 6 and 12
  The HB is a physician-rated system based on criteria of resting appearance, facial movements, and synkinesis that categorizes facial function from I (normal) to VI (total paralysis), with options of "Normal", "Mild dysfunction", "Moderate dysfunction", "Moderately severe dysfunction",", "Severe dysfunction" or "Total paralysis". The prognoses of grade 3 or higher were abnormal.

SECONDARY OUTCOMES:
Sunnybrook Facial Grading Scale (SB Grading) | Baseline, month 3, 6 and 12
  The Sunnybrook Facial Grading Scale was used because of its international recognition and because it allowed a separate classification of the degree of synkinesis. The SB Grading is divided into three subscales of resting symmetry (Eye and Mouth range from 0 to 1, Cheek ranges from 0 to 2), symmetry of voluntary movement (ranges from 1 to 5), and synkinesis (ranges from 0 to 3). The three subscores are used to calculate a composite score (ranges from 0 to 100).
Facial Clinimetric Evaluation Scale (FaCE Scale) | Baseline, month 3, 6 and 12
  FaCE is 15-items, self-reported questionnaire that used to assess facial impairment and disability after facial paralysis. It includes six independent domains: social function, facial movement, facial comfort, oral function, eye comfort, and lacrimal control. the total scores range from 0 (worst) to 100 (best).
Electroneuronography (ENoG) | Baseline, month 3, 6 and 12
  The goal of the Electroneurography (ENoG) testing is to measure the amount of neural degradation that has occurred distal to the site of facial nerve injury by measuring the muscle response to an electrical stimulus. The testing of ENoG involves recording the compound muscle action potential (CAMP) of the mimetic muscles, including Orbicularis oculi and Orbicularis oris muscle. ENoG is performed first on the healthy side of the face and then on the affected side. Nerve damage or nerve fiber degeneration leads to a decrease or loss of the CAMP. The amplitude of the CAMP on the affected side is compared to the CAMP of the healthy side and expressed as percent (amplitude of the paralyzed side divided by the amplitude of the normal side). A side difference of 30% or bigger is considered pathologic.
Electromyography (EMG) | Baseline, month 3, 6 and 12
  EMG is an electrophysiologic measures that indirectly quantify facial nerve function by recording motor unit action potentials (MUAPs) in the muscle of Frontalis muscle. MUAPs are the spikes in electrical activity generated when a motor unit fires. A motor unit consists of a motor neuron and the corresponding muscle fibers innervated by the neuron.
Blink Reflex | Baseline, month 3, 6 and 12
  The blink reflex test is to measures the facial nerve since the blink reflex delivers information on facial nerve function with normal trigeminal function. Blink reflex testing involves electrical stimulation of the supraorbital nerve on the affected side combined with a 2-channel simultaneous sEMG recording from both orbicularis oculi muscles. The exit of the supraorbital nerve in the supraorbital foramen is palpated on the rim of the orbit. Stimulation with 10-20 mA and 0.2 ms duration is used to produce a constant reflex. In blink reflex testing, two responses, R1 and R2, are analyzed. R1 is the fast ipsilateral response of the orbicularis oculi muscle with a latency of about 10-12 ms. The second bilateral response R2 has a latency of about 30-41 ms. The R2 latency differences between both sides higher than 5-8 ms is considered pathologic.

CONTACTS AND LOCATIONS:
Locations (1):
- China Beijing TongRen Hospital, Capital Medical University Beijing, China, Beijing, Beijing Municipality, China